CLINICAL TRIAL: NCT03973632
Title: A Phase I, Open-label, Single-center, Crossover Design of Food-effect Study of SH-1028 Tablets in Healthy Subjects
Brief Title: Pharmacokinetic Study of SH-1028 Tablets in Healthy Subjects Under Fasting and Fed Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHC013-I-03
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — SH-1028

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Fasting at last 10h before taking 200mg（two pills）of SH-1028 tablets on Day 1 of cycle 1，Feeding with high-fat diet within 30 minutes before taking 200mg（two pills）of SH-1028 tablets on Day 1 of cycle 2. Each cycle is 4 days with a 3-days interval.
  Interventions: Drug: SH-1028 Tablets
- Group B (Experimental): Feeding with high-fat diet within 30 minutes before taking 200mg（two pills）of SH-1028 tablets on Day 1 of cycle 1，Fasting at last 10h before taking 200mg（two pills） of SH-1028 tablets on Day 1 of cycle 2. Each cycle is 4 days with a 3-days interval.
  Interventions: Drug: SH-1028 Tablets

INTERVENTIONS:
Drug: SH-1028 Tablets — 200mg of SH-1028 Tablets, orally once every cycle.

SUMMARY:
To evaluate the food-effect of SH-1028 Tablets by pharmacokinetics in healthy subjects under fasting and fed conditions.

DETAILED DESCRIPTION:
By analyzing safety and pharmacokinetics of SH-1028 Tablets in healthy subjects, pharmacokinetic characteristic will be evaluated mainly under fasting and fed conditions.Safety including AE/SAE is also a significant secondary objective.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Subject with acceptable laboratory results.
2. BMI between 19 and 26; Weight between 50 and 80 kg
3. Not allowed to smoke or drink during the trial.
4. Subject should be willing to contracept during the study and until 6 months after completion of study.

Exclusion Criteria:

1. Any clinically relevant abnormalities in physical examination, vital signs, hematology, clinical chemistry, urinalysis or ECG at baseline in the opinion of the Investigator.
2. History of severe allergy/hypersensitivity or or ongoing allergy/hypersensitivity
3. Addicted to smoking and drinking.
4. Hemorrhage over 200mL in 3 months before the trial.
5. Other conditions not suitable for trial, by judgement of investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic of SH-1028 Tablets by assessment of the area under the plasma concentration-time curve from zero to infinity (AUC) | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2(Each cycle is 4 days with a 3-days interval).
Pharmacokinetic of SH-1028 Tablets by assessment of the area under the plasma concentration-time curve from zero to last measurable concentration [AUC(0-t)] | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Every cycle is 4 days with a 3-days interval).
Pharmacokinetic of SH-1028 Tablets by assessment of time to Cmax (tmax) | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Every cycle is 4 days with a 3-days interval).

SECONDARY OUTCOMES:
Adverse event（AE）rate and serious adverse event（SAE）rate | From signing of informed consent to ending of the trial, about 25 days.
Pharmacokinetic of SH-1028 Tablets by assessment of maximum plasma concentration (Cmax) | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Each cycle is 4 days with a 3-days interval).
Pharmacokinetic of SH-1028 Tablets by assessment of terminal rate constant (λz) [ | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Each cycle is 4 days with a 3-days interval).
Pharmacokinetic of SH-1028 Tablets by assessment of Terminal half life (t1/2） | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Each cycle is 4 days with a 3-days interval).
Pharmacokinetic of SH-1028 Tablets by assessment of apparent plasma clearance (CL/F) | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Each cycle is 4 days with a 3-days interval).
Pharmacokinetic of SH-1028 Tablets by assessment of apparent volume of distribution (Vz/F) | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Each cycle is 4 days with a 3-days interval).
Pharmacokinetic of SH-1028 Tablets by assessment of Mean Residence Time（MRT） | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Each cycle is 4 days with a 3-days interval).
Pharmacokinetic of SH-1028 Tablets by assessment of AUC[%Extrap obs],the rate of AUC(t-∞) to AUC | Blood samples are collected pre dose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours post dose on first day of cycle 1 and 2 (Each cycle is 4 days with a 3-days interval).

IPD SHARING:
Plan to Share IPD: No